CLINICAL TRIAL: NCT00521131
Title: Evaluation of Efficacy, Using the Number of Comfortable Days and the Safety of Levocetirizine Dihydrochloride, Administered Once Daily in the Evening for 30 Days, to Subjects Suffering From Perennial Allergic Rhinitis to House Dust Mites
Brief Title: Evaluation of Efficacy and Safety of Levocetirizine to Subjects With Perennial Allergic Rhinitis to House Dust Mites
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A00333
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2009-09

CONDITIONS: Rhinitis; Allergic; Perennial
Keywords: Levocetirizine dihydrochloride; Xyzal tablets
MeSH Terms: conditions — Rhinitis | interventions — levocetirizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Levocetirizine dihydrochloride

SUMMARY:
Evaluation of Efficacy and Safety of Levocetirizine to Subjects With Perennial Allergic Rhinitis to House Dust Mites

ELIGIBILITY:
Inclusion Criteria:

* male or female ≥ 12 years
* suffering from a perennial allergic rhinitis to house dust mites for at least 2 years
* positive skin test or positive Radio-Allergo-Sorbent-Test for house dust mites
* the mean of the T4SS evaluated in the evening over the last 24 hours of the selection period was ≥ 5

Exclusion Criteria:

* seasonal allergic rhinitis likely to change significantly the symptoms of the subject
* an ear, nose or throat (ENT) infection during the two weeks preceding initial visit
* asthma requiring corticosteroid treatment
* atopic dermatitis or urticaria requiring an antihistamine treatment or the administration of oral or topical corticosteroids
* associated ENT disease

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2002-09; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Number of comfortable days, as assessed by the subject | 30 days

SECONDARY OUTCOMES:
Sum of 4 and 5 rhinitis symptoms and safety | Week 1 and over 30 days

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma